CLINICAL TRIAL: NCT04640207
Title: Prospective, Single-Center, Open-Label Study to Evaluate the Efficacy of the Alma Hybrid System for New Approach of Facial Skin Treatment With Minimal Downtime
Brief Title: The Efficacy of the Alma Hybrid System for a New Approach of Facial Skin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-Hyb-Pro-20-011
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Facial skin treatment (Experimental): Facial skin treatment using the Alma Hybrid system.
  Interventions: Device: Facial skin treatment

INTERVENTIONS:
Device: Facial skin treatment — Facial skin treatment using the Alma Hybrid system with a unique pattern that includes both ablative and non-ablative wavelengths

SUMMARY:
The study is aimed to evaluate the efficacy of the Alma Hybrid system for a new approach of facial skin treatment, using both ablative and non-ablative wavelengths.

The study will include 20 subjects with mild-moderate photodamaged skin, that will undergo 2 facial skin treatments. Follow up visit to evaluate the efficacy of the treatments will take place 1 and 3 months after the last treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or Female, 35 to 60 years of age, at the time of enrollment
2. Fitzpatrick skin type I-IV
3. Mild-moderate photo damages and wrinkles, with Fitzpatrick-Goldman Wrinkle and Elastosis Score of 3-6

Main Exclusion Criteria:

1. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
2. Heavy smoker (>1 pack of cigarettes a day)
3. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study
4. Previous rejuvenation treatments on the same area, such as chemical peel, dermabrasion, non-ablative or ablative resurfacing procedure, or face-lift with laser or other devices, up to 3 months prior to the enrollment
5. Prior use of collagen, fat injections, or other methods of skin augmentation within the past 12 months.
6. Prior use of Botox in the treatment area within 5 months
7. Infection, dermatitis, rash, or other skin abnormality in the target area
8. History of any disease or condition that could impair wound healing
9. History of keloid formation, hypertrophic scarring, or abnormal/delayed wound healing

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Investigator assessment | 3 month after last treatment
  Investigator assessment of the overall facial skin aesthetic appearance using a 5 point Likert scale (when "1" indicate "not at all improved" and "5" indicates " very much improved"

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Griffin, MD, Principal Investigator — Dermatology Associates of Plymouth Meeting, P.C.
Locations (1):
- Dermatology Associates of Plymouth Meeting, P.C., Plymouth Meeting, Pennsylvania, United States